CLINICAL TRIAL: NCT00988364
Title: Effects of Ezetimibe, Simvastatin, and Vytorin on Reducing L5 in Patients With Metabolic Syndrome
Brief Title: Effects of Ezetimibe, Simvastatin, and Vytorin on Reducing L5 a Subfraction of LDL in Patients With Metabolic Syndrome.
Acronym: Merck-123
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Chu-Huang Chen, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-20169; MK0653A (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; LDL subfraction L5; The reduction of LDL in patients with Metabolic Syndrome; The prevalence of L5 in patients with Metabolic Syndrome; The reduction of L5 in patients with Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Simvastatin; Ezetimibe, Simvastatin Drug Combination; Ezetimibe

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled clinical trial with 4 arms
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ezetimibe (Active Comparator): Randomly chosen participants will receive ezetimibe 10mg daily for 3 months.
  Interventions: Drug: Ezetimibe
- Simvastatin (Active Comparator): Randomly chosen participants will receive Simvastatin 20mg daily for 3 months.
  Interventions: Drug: Simvastatin
- Vytorin (Active Comparator): Randomly chosen participants will receive Vytorin 20/10mg daily for 3 months.
  Interventions: Drug: Vytorin
- Placebo (Placebo Comparator): Randomly chosen participants will receive Placebo tab 1 daily for 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 20mg daily for 3 months.
  Other Names: Zocor
  Arms: Simvastatin
Drug: Vytorin — Vytorin 20/10mg daily for 3 months.
  Other Names: Ezetimibe/Simvastatin
  Arms: Vytorin
Drug: Placebo — Placebo one tablet daily times 3 months.
  Other Names: Control
  Arms: Placebo
Drug: Ezetimibe — Ezetimibe 10mg daily for 3 months.
  Other Names: Zetia
  Arms: Ezetimibe

SUMMARY:
The purpose of this study is:

* To identify the common factor for L5 prevalence in patients with Metabolic Syndrome.
* To determine whether Ezetimibe, Simvastatin, and Vytorin can correct the L5- promoting factor and reduce L5 in Metabolic Syndrome patients.

DETAILED DESCRIPTION:
Epidemiological evidence indicates that metabolic syndrome (MS) is a strong predisposing condition for atherosclerosis. Elevation of plasma low-density lipoprotein (LDL) cholesterol(LDL-C) concentration is the most important risk factor for atherosclerosis; however, LDL-C elevation is not a criterion for metabolic syndrome, raising the question of LDL's role in the syndrome's association with atherosclerosis. L5, a highly electronegative and mildly oxidized LDL subfraction that we recently isolated from hypercholesterolemic human plasma, may provide a key to answering this question. In cultured vascular endothelial cells (EC), L5 inhibits proliferation and induces apoptosis and monocyte-EC adhesion. In our preliminary studies, L5 could also be detected in patients with MS without elevated LDL-C. Because other LDL subfractions were harmless to EC, the presence of MS-L5 prompted us to hypothesize that the atherogenic role of LDL is not solely determined by plasma LDL-C concentration, but more importantly, by its composition. The proposed study is designed to test this hypothesis. The first question we will address is what lipid factor determines the prevalence of L5 in MS.

Subsequently, we will examine whether treatment with selected medicines can effectively reduce L5 in MS patients by correcting the factor favorable for L5 formation.

We are in the process of identifying the active components of L5 to fully characterize the atherogenic role of L5 in MS,. In the current proposal, we focus our interest on the efficacy of Ezetimibe, Simvastatin, and Vytorin in reducing L5 from the plasma of MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet 3 or more of the 5 criteria specified in the ATPIII guidelines will be recruited.
* The 5 criteria are:

  1. abdominal obesity (men>40 inches, women >35 inches);
  2. TG> 150mg/dL;
  3. low HDL-C (men < 40mg/dL, women < 50 mg/dL);
  4. high blood pressure (>or=130/>or=85 mmHg);
  5. fasting glucose > or = 110mg/dL.
* People with different ethnic backgrounds will be included.

Exclusion Criteria:

* symptomatic coronary artery disease
* peripheral vascular disease
* cerebral ischemia (stroke)
* smoking
* hypothyroidism
* kidney diseases
* consumption of antioxidation supplements/drugs or use of lipid-lowering drugs in the last 3 months
* women who are pregnant, nursing, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chu-Huang Chen, M.D., Ph.D., Principal Investigator — Baylor College of Medicine; Christie Ballantyne, M.D., Study Director — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Avogaro P, Cazzolato G, Bittolo-Bon G. Some questions concerning a small, more electronegative LDL circulating in human plasma. Atherosclerosis. 1991 Nov;91(1-2):163-71. doi: 10.1016/0021-9150(91)90198-c. PMID 1811552
- [Background] Ballantyne CM, Houri J, Notarbartolo A, Melani L, Lipka LJ, Suresh R, Sun S, LeBeaut AP, Sager PT, Veltri EP; Ezetimibe Study Group. Effect of ezetimibe coadministered with atorvastatin in 628 patients with primary hypercholesterolemia: a prospective, randomized, double-blind trial. Circulation. 2003 May 20;107(19):2409-15. doi: 10.1161/01.CIR.0000068312.21969.C8. Epub 2003 Apr 28. PMID 12719279
- [Background] Ballantyne CM, Hoogeveen RC, Bang H, Coresh J, Folsom AR, Heiss G, Sharrett AR. Lipoprotein-associated phospholipase A2, high-sensitivity C-reactive protein, and risk for incident coronary heart disease in middle-aged men and women in the Atherosclerosis Risk in Communities (ARIC) study. Circulation. 2004 Feb 24;109(7):837-42. doi: 10.1161/01.CIR.0000116763.91992.F1. Epub 2004 Feb 2. PMID 14757686
- [Background] Chan DC, Watts GF, Barrett PH, Mamo JC, Redgrave TG. Markers of triglyceride-rich lipoprotein remnant metabolism in visceral obesity. Clin Chem. 2002 Feb;48(2):278-83. PMID 11805008
- [Background] Chen CH, Jiang T, Yang JH, Jiang W, Lu J, Marathe GK, Pownall HJ, Ballantyne CM, McIntyre TM, Henry PD, Yang CY. Low-density lipoprotein in hypercholesterolemic human plasma induces vascular endothelial cell apoptosis by inhibiting fibroblast growth factor 2 transcription. Circulation. 2003 Apr 29;107(16):2102-8. doi: 10.1161/01.CIR.0000065220.70220.F7. Epub 2003 Apr 14. PMID 12695302
- [Background] Chen CH, Pace PW, Karakoc ND, Lu J, Chen HH, Henry PD, Pownall HJ Foreyt JP, Ballantyne CM, Yang CY. Effective reduction of novel atherogenic LDL subfraction by atorvastatin in patients with hypercholesteremia. J AM Coll Cardiol. 2004:43(suppl A):486A (Abstract)
- [Background] Chappey B, Myara I, Benoit MO, Maziere C, Maziere JC, Moatti N. Characteristics of ten charge-differing subfractions isolated from human native low-density lipoproteins (LDL). No evidence of peroxidative modifications. Biochim Biophys Acta. 1995 Dec 7;1259(3):261-70. doi: 10.1016/0005-2760(95)00172-7. PMID 8541333
- [Background] De Castellarnau C, Sanchez-Quesada JL, Benitez S, Rosa R, Caveda L, Vila L, Ordonez-Llanos J. Electronegative LDL from normolipemic subjects induces IL-8 and monocyte chemotactic protein secretion by human endothelial cells. Arterioscler Thromb Vasc Biol. 2000 Oct;20(10):2281-7. doi: 10.1161/01.atv.20.10.2281. PMID 11031216
- [Background] Demuth K, Myara I, Chappey B, Vedie B, Pech-Amsellem MA, Haberland ME, Moatti N. A cytotoxic electronegative LDL subfraction is present in human plasma. Arterioscler Thromb Vasc Biol. 1996 Jun;16(6):773-83. doi: 10.1161/01.atv.16.6.773. PMID 8640405
- [Background] Kleinman Y, Krul ES, Burnes M, Aronson W, Pfleger B, Schonfeld G. Lipolysis of LDL with phospholipase A2 alters the expression of selected apoB-100 epitopes and the interaction of LDL with cells. J Lipid Res. 1988 Jun;29(6):729-43. PMID 2459282
- [Background] La Belle M, Blanche PJ, Krauss RM. Charge properties of low density lipoprotein subclasses. J Lipid Res. 1997 Apr;38(4):690-700. PMID 9144084
- [Background] Lee SJ, Campos H, Moye LA, Sacks FM. LDL containing apolipoprotein CIII is an independent risk factor for coronary events in diabetic patients. Arterioscler Thromb Vasc Biol. 2003 May 1;23(5):853-8. doi: 10.1161/01.ATV.0000066131.01313.EB. Epub 2003 Mar 13. PMID 12637336
- [Background] Libby P. Inflammation in atherosclerosis. Nature. 2002 Dec 19-26;420(6917):868-74. doi: 10.1038/nature01323. PMID 12490960
- [Background] Sanchez-Quesada JL, Benitez S, Ordonez-Llanos J. Electronegative low-density lipoprotein. Curr Opin Lipidol. 2004 Jun;15(3):329-35. doi: 10.1097/00041433-200406000-00014. PMID 15166790
- [Background] Sevanian A, Bittolo-Bon G, Cazzolato G, Hodis H, Hwang J, Zamburlini A, Maiorino M, Ursini F. LDL- is a lipid hydroperoxide-enriched circulating lipoprotein. J Lipid Res. 1997 Mar;38(3):419-28. PMID 9101423
- [Background] Steinberg D. Lewis A. Conner Memorial Lecture. Oxidative modification of LDL and atherogenesis. Circulation. 1997 Feb 18;95(4):1062-71. doi: 10.1161/01.cir.95.4.1062. No abstract available. PMID 9054771
- [Background] Simons L, Tonkon M, Masana L, Maccubbin D, Shah A, Lee M, Gumbiner B. Effects of ezetimibe added to on-going statin therapy on the lipid profile of hypercholesterolemic patients with diabetes mellitus or metabolic syndrome. Curr Med Res Opin. 2004 Sep;20(9):1437-45. doi: 10.1185/030079904x2321. PMID 15383192
- [Background] van Heek M, Austin TM, Farley C, Cook JA, Tetzloff GG, Davis HR. Ezetimibe, a potent cholesterol absorption inhibitor, normalizes combined dyslipidemia in obese hyperinsulinemic hamsters. Diabetes. 2001 Jun;50(6):1330-5. doi: 10.2337/diabetes.50.6.1330. PMID 11375333
- [Background] Yang CY, Raya JL, Chen HH, Chen CH, Abe Y, Pownall HJ, Taylor AA, Smith CV. Isolation, characterization, and functional assessment of oxidatively modified subfractions of circulating low-density lipoproteins. Arterioscler Thromb Vasc Biol. 2003 Jun 1;23(6):1083-90. doi: 10.1161/01.ATV.0000071350.78872.C4. Epub 2003 Apr 10. PMID 12689919
- [Background] Yang CY, Chen HH, Huang MT, Raya JL, Yang JH, Chen CH, Gaubatz JW, Pownall HJ, Taylor AA, Ballantyne CM, Jenniskens FA, Smith CV. Pro-apoptotic low-density lipoprotein subfractions in type II diabetes. Atherosclerosis. 2007 Aug;193(2):283-91. doi: 10.1016/j.atherosclerosis.2006.08.059. Epub 2006 Oct 9. PMID 17030034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 30 enrolled participants, 24 met inclusion criteria and were randomized to treatment.
Groups:
- Ezetimibe: Participants take Ezetimibe 10mg daily for 3 months. N= 6
- Simvastatin: Participants take Simvastatin 20mg daily for 3 months. N=6
- Vytorin: Participants take Vytorin 20/10mg daily for 3 months. N=6
- Placebo: Participants take Placebo tab 1 daily for 3 months. N=6
Period: Overall Study
Arm/Group | Ezetimibe | Simvastatin | Vytorin | Placebo
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ezetimibe: Participants take Ezetimibe 10mg daily for 3 months. N= 6 Ezetimibe: 10mg tablet
- Simvastatin: Participants take Simvastatin 20mg daily for 3 months. N=6 Simvastatin: 20mg tablet
- Vytorin: Participants take Vytorin 20/10mg daily for 3 months. N=6 Vytorin: 20/10mg tablet
- Placebo: Participants take Placebo tab 1 daily for 3 months. N=6 Placebo: 1 tablet
- Total: Total of all reporting groups
Arm/Group | Ezetimibe | Simvastatin | Vytorin | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (4.61) | 49.5 (7.71) | 52.8 (4.22) | 52 (9.01) | 52 (6.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 3 | 3 | 14
  Male | 3 | 1 | 3 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2 | 4
  White | 4 | 2 | 2 | 0 | 8
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 2 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: L5 Concentration in Metabolic Syndrome Patients
Description: Patient's blood samples were collected before treatment. L5 were purified by ultracentrifugation then FPLC. Quantification analysis will indicate the L5 concentration (mg/dL) per group.
Time Frame: 0 months, at the start
Population: all participants assigned to Ezetimibe, Simvastatin, Vytorin and Placebo will receive the corresponding treatment according to the assigned group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ezetimibe | Simvastatin | Vytorin | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
mg/dL | 35.97 (28.87) | 17.8233 (14.4558) | 29.736 (21.143) | 23.1 (18.338)

2. Secondary Outcome: L5 Concentration After Treatment of Ezetimibe, Simvastatin, or Vytorin in Metabolic Syndrome Patients
Description: Patient's blood samples were collected at the corresponding time point for L5 purification. L5 quantification and characterization were investigated with chemical analysis, proteomics and in-vitro cell signaling analysis. Final data analysis will determine total L5 concentration (mg/dL).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ezetimibe | Simvastatin | Vytorin | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
mg/dL | 30.17 (21.66) | 19.19 (19.4648) | 14.17 (16.721) | 15.15 (15.027)

ADVERSE EVENTS:
Time Frame: 3 months later
Description: After 3 months treatment, all participants went through systematic review of any serious adverse events (such as stain-associated muscle symptoms), other adverse events, and all-cause mortality.
Arm/Group | Ezetimibe | Simvastatin | Vytorin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe (N=6) | Simvastatin (N=6) | Vytorin (N=6) | Placebo (N=6)
statin-associated muscle symptoms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No